CLINICAL TRIAL: NCT03237520
Title: Comparing Efficacy of Virtual Reality Therapy With Modified Constraint Induced Movement Therapy (mCIMT) Versus mCIMT Alone, for 5-18 Years Children With Hemiparetic Cerebral Palsy - An Open Label, Randomized Controlled, Superiority Trial
Brief Title: Comparing Virtual Reality Therapy With Modified-CIMT Versus Modified-CIMT Alone in Hemiparetic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRT with CIMT vs CIMT alone
Record Dates: First submitted 2017-07-23; First posted 2017-08-02 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Hemiparesis
MeSH Terms: conditions — Paresis | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: An open labeled, randomized controlled, parallel design, superiority trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be masked to the group allocation and the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Therapy (Experimental): Intervention: Virtual Reality therapy(VRT) reinforcing modified Constraint Induced Movement therapy(mCIMT) VRT will be administered using computer based program. mCIMT will be administered using the physical rehabilitation protocol.
  Interventions: Other: Virtual Reality Therapy
- mCIMT (Active Comparator): Intervention: Modified Constraint Induced Movement Therapy Only mCIMT will be administered using the physical rehabilitation protocol.
  Interventions: Other: mCIMT

INTERVENTIONS:
Other: Virtual Reality Therapy — VRT software and device is developed in collaboration with IIT Delhi using Kinect system. Kinect- motion sensor and computer set up is required. VRT (CIMT in a virtual environment)will be provided for 2 hours at every visit(twice weekly for first 4 weeks, once a week for next 4 weeks). VRT will be provided only during scheduled visits with the same principle as mCIMT. Functional activities like repetition of the tasks and shaping will be performed with the affected hand using VRT and CIMT while the unaffected arm is restrained
  Arms: Virtual Reality Therapy
Other: mCIMT — Modified constraint induced movement therapy will be provided to all children according to predefined protocol.
  Arms: mCIMT

SUMMARY:
This study intends to compare the efficacy of of virtual reality therapy(VRT) with modified constraint induced movement therapy(mCIMT) versus modified constraint induced movement therapy alone for children with hemiparetic cerebral palsy aged >/= 5-18 years, in improving the upper limb functions, as measured by the QUEST (Quality of Upper Extremity Skill Test score) over 3 months of intervention.

DETAILED DESCRIPTION:
Sample size: Based on the previous studies, on CIMT in hemiparetic CP children using QUEST scores,

* Anticipated increase in total QUEST scores at 2 months in the mCIMT group:

  10 + 5(mean + SD)
* Anticipated increase in total QUEST scores at 2 months in the mCIMT+ VRT group:

  15 + 5(mean + SD)
* Alpha error= 5%
* Power= 80%
* Calculated sample size : 23 children in each group
* Considering loss due to attrition of roughly 25%,investigators would enroll 30 children in each of the two groups.
* At least 10 children in each group will be analyzed with baseline and follow up fMRI and DTI. These children in each group will be selected through systematic sampling method.

Method:

* Block randomization in 1:1 ratio with variable block size will be done using computer generated random numbers. These will be generated by the person not involved in the trial. Subjects will be randomized to

  * mCIMT + VRT
  * mCIMT alone
* Each random number will be kept in an opaque sealed envelope and will be opened only at the time of enrollment of the study subjects.Principal investigator will then enroll the participants, and will assign the participants to interventions. After obtaining informed consent from parents, and assent from the children participating in the trial(whenever possible), of hemiparetic cerebral palsy, subjects will be enrolled in the study as per the inclusion and exclusion criteria. Details for each patient will be recorded in a structured proforma

The total study duration will be 3 months, of which 2 months of supervised intervention will be given.Home based therapy will be continued all through the 3 months of intervention in both the groups.

* Functional assessment of the upper limbs will be done using QUEST/Nine Hole Peg Board Test/ Hand Held Dynamometer and quality of life by cerebral palsy quality of life(CP-QOL)- child scale. Baseline fMRI(Functional Magnetic Resonance Imaging) and DTI(Diffusion Tensor Imaging) Brain will be performed up to one week before starting intervention.
* Baseline fMRI and DTI will be done in at least 10 children of each group, selected by systematic sampling method within each group.
* mCIMT+ VRT program will be initiated within one week of baseline assessment, at the institute(Department of PMR). There will be 12 visits over the duration of intervention for supervised sessions, in each group. It would be twice weekly for 4 weeks followed by once a week for next 4 weeks. Parents will be advised regarding the therapy to be provided at home on these visits. Compliance log will be provided to them at the first visit
* Compliance log will be checked on each subsequent visit; reinforcement will be provided; video records of one session per week of each item of mCIMT done at home will also be reviewed. Those following regimen for <70 % of the total time recommended for mCIMT each day for at least 21 out of 28 days will be considered to be poorly compliant. Those following regimen for >80% of the total time recommended for mCIMT each day for at least 21 out of 28 days will be considered to have compliance. Those following the regimen for 80-90% of the total time recommended for mCIMT each day for at least 21 out of 28 days will be considered to have fair compliance.Those following the regimen for >90% of the total time recommended for mCIMT each day for at least 21 out of 28 days will be considered to have good compliance.[All children(both with good and poor compliance), will be included in the intention to treat analysis]

CIMT(Control group and intervention group) :

• Sling will be applied to the unaffected arm, as a restraint (sling will be provided free of cost). mCIMT will be performed for 2 hours per session during the scheduled visits(in the control group) and 2 hours every day at home(by both the groups). Functional activities will be carried out by the affected, unrestrained arm under supervision. Repetitive activities and shaping will be practiced. mCIMT will be provided by trained occupational therapist, first investigator and with the caregiver's participation and would be tailor made to each patient. At each visit, the methodology followed at home will be reviewed (log books with/without video records). Reinforcement will be provided at each visit regarding subsequent therapy to be done at home.

VRT(Intervention group only):

* VRT software and device is developed in collaboration with IIT Delhi using Kinect system. Kinect- motion sensor and computer set up is required. VRT (CIMT in a virtual environment)will be provided for 2 hours at every visit(twice weekly for first 4 weeks, once a week for next 4 weeks). VRT will be provided only during scheduled visits with the same principle as mCIMT. Functional activities like repetition of the tasks and shaping will be performed with the affected hand using VRT and CIMT while the unaffected arm is restrained. At home, 2 hours of modified CIMT will be given daily, as for the control group. At each visit, the methodology of CIMT followed at home is reviewed (log books with/without video records). Reinforcement will be provided at each visit regarding subsequent therapy to be done at home
* FMRI and DTI will be done within 1 week of completion of 08 weeks of intervention in all those children who have had a baseline fMRI/DTI.
* After 8 weeks of intervention, children will be followed up again at the end of 12 weeks from the baseline. They will be asked to continue mCIMT daily for 2 hours at home and maintain the daily logs during this period. At this visit, all clinical assessments will be repeated
* Outcome assessors will be blinded to the study subject's group allocation.
* Data will be recorded in a pre-designed proforma and managed in an excel spread sheet.All the entries will be checked for any possible key board errors. Statistical analysis will be done using Stata 14.0 statistical software.
* Intention to treat analysis and per protocol analysis will be done
* Categorical variables will be summarized by frequency (%) and test of proportions will be used to compare the proportions between the two groups. Quantitative variables will be assessed for approximate normal distribution and these will be denoted as mean+SD or median (Interquartile range/min-max), as appropriate.Student's t test/ Wilcoxon rank sum test will be used to compare the mean value between the two groups at the end of the intervention and at the end of 3 months. In case of any imbalance at the baseline, analysis of covariance(ANCOVA) will be used to compute adjusted mean of the outcome variables bet the two groups and the corresponding effect size(95%CI).In this study p value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged >5-18 years
2. Children with hemiparetic cerebral palsy * (both perinatal and postnatal acquired brain injury)
3. Intelligence quotient >70 (Binet Kamat Test/Malin's Intelligence Scale for Children)
4. Modified Ashworth scoring 1-3 for affected limb
5. Can sit independently or with support (Gross Motor Functional Classification System stage: 1-4 and Manual Ability Classification System stage: 1-3)
6. Preserved vision and hearing (with or without correction)

Exclusion Criteria:

1. Uncontrolled epilepsy as defined by seizure frequency >1/month for preceding 3 months
2. Severe concurrent illness or diseases not associated with CP or unstable medical conditions like pneumonia
3. Genetic or syndromic associations
4. Children diagnosed with autistic spectrum disorders
5. Modified Ashworth scale score more than 3 at shoulder/elbow /wrist
6. Contractures of the affected limb
7. Severe movement disorder like dystonia, choreo-athetosis or ballismus interfering with purposeful limb movement
8. Any congenital brain malformation detected on conventional MRI brain
9. Recent orthopedic surgery/cast/splint in the affected limb
10. Botulinum toxin/phenol blocking in the affected limb in the past 6 months or are planning to receive in the study period
11. Those receiving tone modifying agents in week before enrollment(Tizanidine,baclofen,benzodiazepines,dantrolene)
12. Any contraindications for MRI - examples- presence of pacemaker, metallic implant

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
8 weeks of VRT with mCIMT versus mCIMT alone | Within 1 week of completing 8 weeks, from the beginning of intervention
  The primary objective is to evaluate and compare the efficacy of 8 weeks of modified constraint induced movement therapy (mCIMT) reinforced with virtual reality therapy(VRT) with modified constraint induced movement therapy alone, in improving the upper limb function in >5-18 years old children with hemiparetic cerebral palsy, by using the QUEST scoring(Quality Of Upper Extremity Skill Test Score) in the two groups.

SECONDARY OUTCOMES:
To compare the improvement in the sub domains(dissociated movements, grasp, protective extension and weight bearing) of QUEST score between the 2 groups | Within 1 week of completing 8 weeks, from the beginning of intervention
  QUEST is the Quality Of Upper Extremity Skill Test. It assesses quality of the dissociated movements, grasp, weight bearing and protective extension. In each group at the end of 8 weeks the QUEST score will be chronicled for each of the domains and compared between the intervention and control group.
Comparing the improvement in speed of movements between 2 groups | Within 1 week of completing 8 weeks,from the beginning of intervention
  This will be assessed using the nine hole peg board. The difference in change in mean time to complete the nine hole peg board will be compared between the two groups.
Comparing the improvement in muscle strength between 2 groups | Within 1 week of completing 8 weeks,from the beginning of intervention
  The muscle strength will be assessed by hand held dynamometer. The change in muscle strength measured in pounds by hand held dynamometer will be compared between two groups.
Functional Magnetic Resonance Imaging(fMRI) in the 2 groups | Upto 1 week before starting mCIMT+ VRT program and within 1 week of completing 08 weeks, from the beginning of the intervention
  To describe functional magnetic resonance imaging(fMRI) changes in a pre-defined motor paradigm of the paretic upper limb in terms of changes in BOLD(Blood Level Oxygen Dependent) cluster activation of ipsilesional (contralteral *) somatosensory cortex; laterality Index of Broadmann Area 4 (BA4) and Broadman area 6 (BA6), and ipsilateral cerebellum activation ratio during the motor task performance of the paretic upper limb in fMRI Brain in both the groups
fMRI changes copared with clinical improvement in 2 groups before and after intervention | Upto 1 week before starting mCIMT+ VRT program and within 1 week of completing 08 weeks, from the beginning of the intervention
  This is done by comparing changes in fMRI brain in terms of BOLD cluster activation of contralateral and ipsilateral somatosensory cortex with clinical assessment of upper limb function in terms of QUEST score between the two groups
DTI(Diffusion Tensor Imaging) changes compared with clinical improvement in 2 groups before and after intervention | Upto 1 week before starting mCIMT+ VRT program and within 1 week of completing 08 weeks, from the beginning of the intervention
  This is done by comparing changes in diffusion tensor imaging findings in terms of fractional anisotropy value of the lesion with clinical assessment of upper limb function in terms of QUEST scores between the two groups
Diffusion Tensor Imaging changes in 2 groups | Upto 1 week before starting mCIMT+ VRT program and within 1 week of completing 08 weeks, from the beginning of the intervention
  To describe changes in Diffusion Tensor Imaging findings in terms of fractional anisotropy value of the lesion between the two groups(performed at baseline, and within one week of completion of 8 weeks of intervention)
Sustained improvement | Baseline and at 12 weeks of intervention
  This is done by assessing the difference in change in total QUEST scores at baseline and at 12 weeks of intervention, between the intervention and the control groups, and assessing the persistence of improvement, 4 weeks after stopping supervised intervention.
Quality of life improvement | At the end of 8 weeks, from the beginning of intervention
  Cerebral Palsy- Quality Of Life scale for children(CP-QOL child) will be applied at baseline and at 8 weeks of intervention. Difference in change in CP-QOL scores at baseline and at 8 weeks of intervention will be compared between two groups.
Compliance | At the end of 8 weeks, from the beginning of intervention
  Parents will be asked to maintain daily activity monitoring log. The compliance in two groups will be assessed based on this log.